CLINICAL TRIAL: NCT01033539
Title: To Demonstrate That Lactobacillus Reuteri ATCC PTA 4659 Survives Passage Through the Gastrointestinal Tract of Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Good Food Practice, Sweden (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: CSP U-08-008 BSS
Record Dates: First submitted 2009-12-15; First posted 2009-12-16 (Estimated); Last update posted 2012-03-29 (Estimated); Status verified 2012-03

CONDITIONS: Recovery of Lactobacillus Reuteri ATCC PTA 4659; The Safety of Lactobacillus Reuteri ATCC PTA 4659
Keywords: Survive; safety; lactobacillus Reuteri

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo control (Active Comparator): Placebo control without probiotics ATCC PTA 4659
  Interventions: Other: Probiotic strain ATCC PTA 4659
- ATCC PTA 4659 Low dose (Active Comparator)
  Interventions: Other: Probiotic strain ATCC PTA 4659
- ATCC PTA 4659 high dose (Active Comparator)
  Interventions: Other: Probiotic strain ATCC PTA 4659

INTERVENTIONS:
Other: Probiotic strain ATCC PTA 4659 — Placebo control containing no probiotic strain of ATCC PTA 4659 High dose of ATCC PTA 4659 1*10 10 CFU/bag Low dose of ATCC PTA 4659 1*10 8 CFU/bag
  Other Names: ATCC PTA 4659

SUMMARY:
The purpose of this study is to determine the effects of a sachet containing Lactobacillus Reuteri ATCC PTA 4659 on the recovery of live Lactobacillus reuteri in fecal samples after 7, 14 and 28 days supplementation as well as 14 days wash out compared to the same sachet without the probiotic bacteria as placebo control.

DETAILED DESCRIPTION:
This study is the first to investigate the relative colonisation of the human GI tract by L Reuteri ATCC PTA 4659. Simple demonstration that they survive passage is the first step in development of potential new probiotics, which is necessary before these strains can be considered for continued testing in probiotic food matrices. The aim of this study will evaluate the safety and tolerability of Lactobacillus Reuteri in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Age 18-65 years
* BMI 19-33
* Hb 120 g/women 130 g/l for men
* Healthy assessed by screening tests and physical examination
* Signed informed consent and bio bank consent

Exclusion Criteria:

* Participation in a clinical study within 90 days prior screening use of antibiotics 2 weeks before baseline
* Pregnant or lactating

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-11; Primary Completion 2010-04 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Change form baseline to day 28 on treatment in level of live Lactobacillus Reuteri ATC PTA 4659 in faecal material. | Nov 2009-April2010

CONTACTS AND LOCATIONS:
Overall Officials: Birgitta E Sundberg, PhD, Principal Investigator — Good Food Practice, Uppsala, Sweden
Locations (1):
- Good Food Practice, Uppsala, Uppsala County, Sweden

REFERENCES:
- [Derived] Sendelius M, Axelsson J, Liu P, Roos S. Genomic, phenotypic, and clinical safety of Limosilactobacillus reuteri ATCC PTA 4659. J Ind Microbiol Biotechnol. 2023 Feb 17;50(1):kuad041. doi: 10.1093/jimb/kuad041. PMID 37974056